CLINICAL TRIAL: NCT04202107
Title: Development and Evaluation of a Semi-quantitative Food Frequency Questionnaire for Use in Urban and Rural Communities of Rwanda
Brief Title: Dietary Assessment in Rwanda - Food Frequency Questionnaire
Acronym: FFQ Rwanda
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: University of Rwanda (Other); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Responsible Party: Sponsor
Other Study IDs: EC/2019/1578
Record Dates: First submitted 2019-11-27; First posted 2019-12-17 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Dietary Assessment
Keywords: Dietary assessment; Food Frequency Questionnaire; multi-pass 24 hour food recall; semi-quantitative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urban: Men and women between 18 and 49 years of age living in the selected urban communities in Rwanda and who are familiar with the diet.
  Participants in this study should be acquainted with cooking practices to be able to cite all the ingredients that are used in the preparation of the dishes/ meals
  Interventions: Other: Food Frequency Questionnaire; Other: 24 Hour food recall
- Rural: Men and women between 18 and 49 years of age living in the selected urban communities in Rwanda and who are familiar with the diet.
  Participants in this study should be acquainted with cooking practices to be able to cite all the ingredients that are used in the preparation of the dishes/ meals
  Interventions: Other: Food Frequency Questionnaire; Other: 24 Hour food recall

INTERVENTIONS:
Other: Food Frequency Questionnaire — Food frequency questionnaires (FFQs) are a common method for measuring dietary intake in large epidemiological studies, in particular in low literacy settings were diaries and food history would not be viable.
Other: 24 Hour food recall — Standardized and validated approach of collecting all foods, beverages, and supplements consumed during the past 24 hours

SUMMARY:
The burden of non-communicable diseases (NCDs) in Rwanda is adding to the health burden in the country which is facing the nutritional transition and the double burden of malnutrition. Diet is an established risk factor in NCDs, hence the importance to assess accurately the changes in dietary habits occurring in the population. The objective is to develop and validate a food frequency questionnaire in Rwanda.

DETAILED DESCRIPTION:
In many developing countries, including Rwanda, the lack of developed and validated questionnaires is among major challenges for dietary assessment in nutritional surveys. Questionnaires are mostly borrowed from other communities. This can increase the error range due to low adaptation to local context, especially when they are not validated and may not have similar objectives. One Food Frequency Questionnaire (FFQ) does not capture dietary history in two different countries or regions, unless their diets are similar. Besides, the diet changes with time, where new foods are introduced in diet and others may disappear. In Rwanda, one FFQ has been developed to cover only the eastern part of the country, but none for the entire country (Cade et al., 2001; FAO, 2018). It is then very important to develop and validate an update and general FFQ that can be used across the country to measure the dietary intake to have a better interpretation of the study findings from the Rwandan context.

The overall objective is to develop and validate a semi-quantitative FFQ that can be used to assess the food and nutrient intake in urban and rural communities of Rwanda.

Specific objectives include:

1. To collect data on diet intake of selected participants by using a 24-H recall questionnaire that includes pictures on the approximate quantities consumed in each occasion.
2. To develop a list of food items from commonly consumed food by study participants using the compiled 24-h recall questionnaire to use for an FFQ development. Additionally, an open question format to collect information on foods consumed during social gathering and festivals will be used to include unreported foods. FFQ shall include additionally the food portion size, and the frequency of intake over a reference period of one year.
3. To assess the accuracy of the developed FFQ in estimating energy and nutrient intake using the 24-H dietary recall as a benchmark of accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Permanent residence of the selected urban or rural villages
* Holding a valid health insurance card
* Aged between 18 and 49 years
* Signing informed consent form
* Familiar with the diet and cooking practices
* Registration in city demographic system, since study participants will be selected from population registration cards at village level,
* Accept enumerators for home visit and data collection for one year

Exclusion Criteria:

* Mental disorders such as clinically diagnosed depression, anxiety disorders, eating disorders and addictive behaviors

Ages: 18 Years to 49 Years | Sex: All
Age Groups: Adult
Study Population: In total, 100 participants will be selected from 100 households (one per household) in urban villages (mainly in Kigali) and the same number of participants from rural communities of Rwanda will be recruited in the validation study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Median proportion of energy intake from carbohydrates assessed by the 24 hour recalls | One year
  Median proportion of energy intake from carbohydrates (starch from grains and tubers such as corn, pasta, rice, potatoes, breads), natural sugars from fruits and juices, and added sugars found in soft drinks, candy, fruit drinks, and desserts) assessed by the 24 hour recalls Adults should get 45 percent to 65 percent of their calories from carbohydrates
Median proportion of energy intake from carbohydrates assessed by the Food Frequency Questionnaire | One year
  Median proportion of energy intake from carbohydrates (starch from grains and tubers such as corn, pasta, rice, potatoes, breads), natural sugars from fruits and juices, and added sugars found in soft drinks, candy, fruit drinks, and desserts) assessed by the Food Frequency Questionnaire.
  Adults should get 45 percent to 65 percent of their calories from carbohydrates
Median proportion of energy intake from fat assessed by the 24 hour recalls | One year
  Median proportion of energy intake from fat (Butter, margarine, vegetable oils, whole milk, visible fat on meat and poultry products, invisible fat in fish, shellfish, some plant products such as seeds and nuts, and bakery products) assessed by the 24 hour recalls.
  Adults should get 20 percent to 35 percent of their calories from fat
Median proportion of energy intake from fat assessed by the Food Frequency Questionnaire | One year
  Median proportion of energy intake from fat (Butter, margarine, vegetable oils, whole milk, visible fat on meat and poultry products, invisible fat in fish, shellfish, some plant products such as seeds and nuts, and bakery products) assessed by the Food Frequency Questionnaire.
  Adults should get 20 percent to 35 percent of their calories from fat
Median proportion of energy intake from proteins assessed by the 24 hour recalls | One year
  Median proportion of energy intake from proteins (from animal sources, such as meat, poultry, fish, eggs, milk, cheese, and yogurt; and proteins from plants, legumes, grains, nuts, seeds, and vegetables) assessed by the 24 hour recalls.
  Adults should get 10 to 35 percent of their calories from protein
Median proportion of energy intake from proteins assessed by the Food Frequency Questionnaire | One year
  Median proportion of energy intake from proteins (from animal sources, such as meat, poultry, fish, eggs, milk, cheese, and yogurt; and proteins from plants, legumes, grains, nuts, seeds, and vegetables) assessed by the Food Frequency Questionnaire.
  Adults should get 10 to 35 percent of their calories from protein
Median daily intake of fibers assessed by the 24 hour recalls | One year
  Median daily intake of fibers (in gram; Includes dietary fiber naturally present in grains, such as found in oats, wheat, or unmilled rice; and functional fiber synthesized or isolated from plants or animals) assessed by the 24 hour recalls.
  The recommended intake for total fiber for adults 50 years and younger is set at 38 grams for men and 25 grams for women
Median daily intake of fibers assessed by the Food Frequency Questionnaire | One year
  Median daily intake of fibers (in gram; Includes dietary fiber naturally present in grains, such as found in oats, wheat, or unmilled rice; and functional fiber synthesized or isolated from plants or animals) assessed by the Food Frequency Questionnaire.
  The recommended intake for total fiber for adults 50 years and younger is set at 38 grams for men and 25 grams for women

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan De Henauw, Md. PhD, Principal Investigator — University Ghent; Souheila Abbeddou, MSc. PhD, Principal Investigator — UGent; Jerome Some, Md. PhD, Principal Investigator — Institut de Recherche en Sciences de la Sante, Ouagadougou, Burkina Faso; Hilda Vasanthakaalam, PhD, Principal Investigator — University of Rwanda
Locations (1):
- University of Rwanda, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowen L, Bharathi AV, Kinra S, Destavola B, Ness A, Ebrahim S. Development and evaluation of a semi-quantitative food frequency questionnaire for use in urban and rural India. Asia Pac J Clin Nutr. 2012;21(3):355-60. PMID 22705424
- [Background] Cade J, Thompson R, Burley V, Warm D. Development, validation and utilisation of food-frequency questionnaires - a review. Public Health Nutr. 2002 Aug;5(4):567-87. doi: 10.1079/PHN2001318. PMID 12186666
- [Background] Aglago EK, Landais E, Nicolas G, Margetts B, Leclercq C, Allemand P, Aderibigbe O, Agueh VD, Amuna P, Annor GA, El Ati J, Coates J, Colaiezzi B, Compaore E, Delisle H, Faber M, Fungo R, Gouado I, El Hamdouchi A, Hounkpatin WA, Konan AG, Labzizi S, Ledo J, Mahachi C, Maruapula SD, Mathe N, Mbabazi M, Mirembe MW, Mizehoun-Adissoda C, Nzi CD, Pisa PT, El Rhazi K, Zotor F, Slimani N. Evaluation of the international standardized 24-h dietary recall methodology (GloboDiet) for potential application in research and surveillance within African settings. Global Health. 2017 Jun 19;13(1):35. doi: 10.1186/s12992-017-0260-6. PMID 28629424
- [Background] Shridhar K, Satija A, Dhillon PK, Agrawal S, Gupta R, Bowen L, Kinra S, Bharathi AV, Prabhakaran D, Srinath Reddy K, Ebrahim S; Indian Migration Study group. Association between empirically derived dietary patterns with blood lipids, fasting blood glucose and blood pressure in adults - the India migration study. Nutr J. 2018 Feb 8;17(1):15. doi: 10.1186/s12937-018-0327-0. PMID 29422041
- See also: The International Dietary Data Expansion (INDDEX) Project — https://inddex.nutrition.tufts.edu/data4diets/data-source/food-frequency-questionnaire-ffq